CLINICAL TRIAL: NCT07158736
Title: Ultrasound-Guided Genicular Nerve Block for Knee Pain in the Emergency Department: A Randomized Controlled Trial
Brief Title: Genicular Nerve Block for Knee Pain in the ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB Protocol #858259
Record Dates: First submitted 2025-07-17; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Knee Pain
MeSH Terms: interventions — Bupivacaine; Adrenal Cortex Hormones; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genicular Nerve Block (Experimental): This arm of patients (17 total) will receive the genicular nerve block for their knee pain.
  Interventions: Procedure: Genicular nerve block with bupivacaine and corticosteroids
- Standard of Care (Active Comparator): This arm of patients (17 total) will receive standard of care analgesia for their knee pain
  Interventions: Other: Standard of Care

INTERVENTIONS:
Procedure: Genicular nerve block with bupivacaine and corticosteroids — genicular nerve block with ideal body-weight dosing of bupivacaine 0.5% with 4 mg dexamethasone
  Arms: Genicular Nerve Block
Other: Standard of Care — This involves standard of care pain relief for patients who do not receive the genicular nerve block for knee pain, such as acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), and opioids.
  Arms: Standard of Care

SUMMARY:
Patient with atraumatic knee pain without a large knee effusion on x-ray will be randomized to receive either a genicular nerve block (GNB) or standard of care in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Atraumatic knee pain
* >17 years age
* X-ray of the knee obtained in the ED
* Initial pain score (numeric rating scale) 5-10

Exclusion Criteria:

* Fracture or dislocation on x-ray
* large knee joint effusion identified on x-ray
* allergy or contraindication to local anesthetics
* History of local anesthetic systemic toxicity after receiving local anesthetics
* Pregnancy
* Incarcerated
* History of knee replacement of affected knee
* Concern for septic joint
* Overlying cellulitis
* Hemodynamic instability
* Altered mental status or inability to consent for procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain level | 1 hour post-enrollment
  Measured by numeric rating scale: 0 (minimum value) - 10 (maximum value)

SECONDARY OUTCOMES:
Difference in Duration of Analgesia | 24 hours
  Patients will be called back to assess their pain levels
Difference in AP-POQ-RED score | 1 hour after enrollment
  9 question survey study, all questions rated on 0 (minimum) - 10 (maximum) scale. Questions include: pain before and after treatment, pain with activities in and out of bed, emotions (anxiety, fear, helplessness), degree of pain relief in the emergency department, satisfaction.
Difference in length of stay in the emergency department | Average 1 hour
  Length of stay in the emergency department is determined from the time the provider first sees the patient to the time the provider discharges the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Shalaby, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Pennsylvania Presbyterian Medical Center, Philadelphia, Pennsylvania
  - HUP Cedar, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT07158736/Prot_000.pdf
  • Informed Consent Form (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT07158736/ICF_001.pdf